CLINICAL TRIAL: NCT07378930
Title: ULTRA-high-risk Surveillance to Avoid Future Events: the ULTRA-SAFE Trial
Acronym: ULTRA-SAFE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, National Taiwan University Hospital, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202511135RINA
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Neoplasms; Colorectal Cancer Prevention; Surveillance Colonoscopy
Keywords: Colonoscopy surveillance; Colorectal cancer prevention; Post-polypectomy surveillance; Fecal immunochemical test
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The trial compares a Standard Arm, which receives routine follow-up colonoscopy at year three, against an Early Screening Group (FIT Arm). In the FIT Arm, participants undergo FIT at years one and two, triggering an earlier colonoscopy if positive. Based on assumptions regarding FIT sensitivity and false-positive rates, the intervention was predicted to reduce the 3-year prevalence of meta-ACRN. The primary endpoint is comparing the recurrence rate of meta-ACRN detected during the third-year surveillance colonoscopy between the two groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care arm (No Intervention): Surveillance colonoscopy performed at third year after initial colonoscopy
- FIT arm (Experimental): Intervention: Early triage using Fecal immunochemical test
  Detailed: Participants in this group will undergo Fecal Immunochemical Testing (FIT) in the first and second years (FIT 1 & 2) following their initial colonoscopy. If FIT 1 is positive, a colonoscopy will be scheduled within three months; regardless of those findings, a surveillance colonoscopy is still required in the third year. If FIT 1 is negative, the patient proceeds to FIT 2 in the second year. A positive FIT 2 likewise triggers a colonoscopy within three months, and a third-year surveillance colonoscopy remains mandatory unless the FIT 2-triggered colonoscopy occurs between 2.5 and 3.5 years after the initial procedure, in which case it fulfills the third-year requirement. If both FIT 1 and FIT 2 are negative, the participant will undergo their scheduled surveillance colonoscopy in the third year.
  Interventions: Diagnostic Test: Early triage using Fecal immunochemical test

INTERVENTIONS:
Diagnostic Test: Early triage using Fecal immunochemical test — Fecal immunochemical test would be provided at first and second year after initial colonoscopy in FIT arm. Those with positive results would be arranged with early surveillance colonoscopy
  Arms: FIT arm

SUMMARY:
The ULTRA-SAFE clinical trial is a prospective, randomized study designed to address the limitations of current "one-size-fits-all" colorectal cancer surveillance guidelines. While international standards recommend a three-year follow-up colonoscopy for all high-risk patients, data suggests that those with multiple advanced adenomas face a significantly higher recurrence risk (20%) compared to those with only low-risk adenomas (9%). To provide more personalized care, the trial compares a Standard Arm (colonoscopy at year three) against a FIT Arm, where participants undergo annual fecal immunochemical testing in years one and two. A positive FIT triggers an earlier colonoscopy, with the goal of reducing the 3-year prevalence of metachronous advanced colorectal neoplasms (meta-ACRN) from 20% to approximately 12.7%. The study has enrolled roughly 940 participants to statistically validate whether this early screening intervention can effectively prevent future malignant events in ultra-high-risk populations.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) prevention is critically dependent on the timely detection and excision of precancerous lesions, particularly advanced adenomas. Advanced adenomas are defined as lesions exceeding one centimeter, or those possessing villous pathology or high-grade dysplasia, representing lesions with high malignant potential. Following the removal of polyps, patients who present with at least three low-risk adenomas or any advanced adenoma are classified as a high-risk population, facing a significantly increased risk of developing metachronous advanced colorectal neoplasms (meta-ACRN), which include metachronous advanced adenoma or CRC, in the future. Current international guidelines recommend that these high-risk individuals undergo follow-up colonoscopy by the third year after initial polyp resection. However, a prior analysis of a multicenter clinical trial in Taiwan revealed substantial diversity in the initial endoscopic presentations among patients with advanced adenomas. This variability in initial findings has been shown to significantly alter the future risk of developing meta-ACRN. For example, for those with multiple advanced adenoma, compared with individuals with 3-10 low-risk adenoma, although they both meet the definition of high-risk population, the risk of 3-year meta-ACRN was 20% and 9%. Therefore, the uniform recommendation for a three-year surveillance follow-up fails to provide personalized advice tailored to this diverse risk profile.

This ULTRA-SAFE clinical trial, which focuses on ULTRA-high-risk Surveillance to Avoid Future Events, is a prospective, randomized controlled study. It aims to determine if implementing early fecal immunochemical testing (FIT) screening can reduce the incidence of meta-ACRN in patients at ultra-high risk. This high-risk group includes individuals who had two or more advanced adenomas detected and removed during their initial colonoscopy. The trial compares a Standard Arm, which receives routine follow-up colonoscopy at year three (where the assumed meta-ACRN prevalence is 20%), against an Early Screening Group (FIT Arm). In the FIT Arm, participants undergo FIT at years one and two, triggering an earlier colonoscopy if positive. Based on assumptions regarding FIT sensitivity and false-positive rates, the intervention was predicted to reduce the 3-year prevalence of meta-ACRN to roughly 12.7%. To statistically detect this difference, a sample size of approximately 402 participants per arm was required. After inflating this number to account for an anticipated 10-15% loss to follow-up, the planned enrollment was set at 470 participants per arm, totaling approximately 940 participants. The primary endpoint is comparing the recurrence rate of meta-ACRN detected during the third-year surveillance colonoscopy between the two groups

ELIGIBILITY:
Inclusion Criteria:

1. Age: Adults aged 40 to 75 years.
2. Initial Colonoscopy Findings: Detection and removal of at least two advanced adenomas during the baseline colonoscopy.
3. Adherence: Willingness to comply with the assigned screening protocol, including fecal immunochemical testing (FIT) and follow-up colonoscopies

Exclusion Criteria:

1. Age: Individuals younger than 40 or older than 75 years.
2. High-Risk Predispositions: Patients with inflammatory bowel disease (IBD), Familial Adenomatous Polyposis (FAP), or a documented hereditary colorectal cancer syndrome (e.g., Lynch syndrome).
3. Cancer History: A history of colorectal cancer (excluding carcinoma in situ).
4. Contraindications: Patients for whom polypectomy is clinically inappropriate or unsafe.
5. Adenoma Count/Type: Failure to meet the requirement of at least two advanced adenomas during the initial colonoscopy.

7.Extensive Low-Risk Lesions: Presence of more than ten low-risk adenomas.

8.Pregnancy: Currently pregnant individuals.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 940 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
3-year incidence of metachronous ACRN | three years after recuitment
  The incidence of metachronous advanced colorectal neoplasm (ACRN: adenoma larger than 1cm OR with villous components OR with high-grade dysplasia OR colorectal cancer) at third-year surveillance colonoscopy in both arms

SECONDARY OUTCOMES:
Overall incidence of metachronous ACRN | 3 years after recruitment
  The incidence of metachronous advanced colorectal neoplasm (adenoma larger than 1cm OR with villous components OR with high-grade dysplasia OR colorectal cancert) at the surveillance colonoscopy at third year in standard-care arm and all surveillance colonoscopy in FIT arm
Overall incidence of metachronous colorectal cancer | three years after recuitment
  The incidence of metachronous colorectal cancer at the surveillance colonoscopy at third year in standard-care arm and all surveillance colonoscopy in FIT arm

IPD SHARING:
Plan to Share IPD: Undecided